CLINICAL TRIAL: NCT00764842
Title: Post-Market Study: The Efficacy of the CLP® Hip
Brief Title: Efficacy of the CLP® Hip - Retrospective
Status: Terminated | Type: Observational
Why Stopped: Enrollment and data collection insufficient to continue study.
Sponsor: Encore Medical, L.P. (Industry)
Responsible Party: Jane M. Jacob Ph.D., DJO Surgical
Other Study IDs: PS - 802
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2011-02

CONDITIONS: Osteoarthritis; Avascular Necrosis; Rheumatoid Arthritis
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CLP Hip
  Interventions: Device: Encore CLP® Hip stem

INTERVENTIONS:
Device: Encore CLP® Hip stem — Subjects with osteoarthritis, rheumatoid arthritis or avascular necrosis of the natural femoral head who have received the Encore CLP® Hip stem and are willing to participate in the study.

SUMMARY:
The purpose of this study is to evaluate the survivorship and efficacy of the Encore CLP® Hip stem in a group of no more than 200 patients from whom data has already been collected.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age or older.
2. Noninflammatory degenerative joint disease including

   * Osteoarthritis of the natural femoral head
   * Avascular necrosis of the natural femoral head
   * Rheumatoid arthritis
3. Correction of functional deformities
4. Femoral fracture
5. Patients must be able and willing to complete all study-related visits.

Exclusion Criteria:

1. Anyone who is under 18 years of age
2. Infection or sepsis
3. Insufficient bone quality which may affect the stability of the implant
4. Muscular, neurological or vascular deficiencies, which compromise the affected extremity
5. Skeletally immature patients and cases where there is a loss of abductor musculature, poor bone stock, poor skin coverage around hip joint which would make the procedure unjustifiable
6. Osteomyelitis
7. Rapid joint destruction or bone absorption apparent on roentgenogram
8. Pathological conditions of the acetabulum which would prevent achieving proper range of motion, appropriate head stability, and/or a well-seated and supported smooth articulation of the head within the acetabulum
9. Alcoholism or other addictions
10. Materials sensitivity
11. Loss of ligamentous structures
12. High levels of physical activity (e.g., competitive sports, heavy physical labor)
13. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who meet the indications for use of the CLP Hip Stem AND who meet the inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2008-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The survivorship and efficacy of the Encore CLP® Hip stem | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: D. Kevin Lester, M.D., Principal Investigator — Center for Excellence
Locations (1):
- Center for Excellence, Fresno, California, United States

REFERENCES:
- See also: Sponsor company home page — http://www.djosurgical.com